CLINICAL TRIAL: NCT04859426
Title: An Open-label, Single-dose, Phase I Study to Assess the Pharmacokinetics and Safety of DBPR108 Tablets in Subjects With Mild, Moderate Hepatic Impairment Compared to the Control Subjects With Normal Hepatic Function
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of DBPR108 in Subjects With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HA1118-CSP-008
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — DBPR108

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mild Hepatic Impairment (Experimental): Subjects will receive a single dose of 100 mg DBPR108.
  Interventions: Drug: DBPR108 tablets
- Moderate Hepatic Impairment (Experimental): Subjects will receive a single dose of 100 mg DBPR108.
  Interventions: Drug: DBPR108 tablets
- Normal hepatic function (Experimental): Subjects will receive a single dose of 100 mg DBPR108.
  Interventions: Drug: DBPR108 tablets

INTERVENTIONS:
Drug: DBPR108 tablets — Drug: DBPR108, tablet, oral
  Other Names: DBPR108

SUMMARY:
This is an open-label, single-dose study to evaluate the pharmacokinetics and safety of DBPR108 in subjects with mild or moderate hepatic impairment (HI) compared to the matched control subjects with normal hepatic function.

DETAILED DESCRIPTION:
DBPR108 is a potent dipeptidylpeptidase-4 inhibitor. The aim of this study is to evaluate the pharmacokinetics and safety of DBPR108 in subjects with mild or moderate hepatic impairment (HI) compared to the matched control subjects with normal hepatic function. This study consists of a screening period (Day -14 to Day -1), a baseline period (Day -1), a treatment period (Day 1 to Day 3), and a follow-up call on Day 6.

Subjects will be enrolled in the following groups:

(A) mild hepatic impairment (Child-Pugh class A, 5-6 points); (B) moderate hepatic impairment (Child-Pugh class B, 7-9 points); (C) control subjects with normal hepatic function will be matched with subjects with HI by weight, age, and sex.

Approximately 8 subjects will be enrolled in each group.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Voluntarily sign the informed consent form, understand the trial procedures, and be willing to comply with all trial procedures and restrictions；
* 18 years to 79 years (inclusive), male or female；
* Male subjects weight ≥50 kg and female subjects weight ≥45 kg. Body mass index (BMI) : 18-30 kg/m2 (inclusive) (BMI= weight (kg)/height 2 (m2))；
* Subjects (including partners) are willing to use effective contraceptives from screening to the 6 months after the last dose administration；

Subjects with HI only:

* Medically stable hepatic impairment on the Child-Pugh Class A (mild) or Child-Pugh Class B (moderate) caused by a primary hepatic disease;
* Not in use of any prescription drug, over-the-counter drug, or herbal medicine within 2 weeks prior to screening, except for the medication necessary for hepatic impairment/ other comorbidities (last more than four weeks in good compliance);

Subjects with normal liver function only:

* Weight, age, and sex must be matched with subjects with HI;
* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) results within normal range;
* Not in use of any prescription drug, over-the-counter drug, or herbal medicine within 2 weeks prior to screening, except for the medication necessary for underlying conditions other than liver disease (last more than four weeks in good compliance);

Exclusion Criteria:

All subjects:

* Subjects who have a history of allergic conditions (such as asthma, urticaria), or have a history of allergy to two or more drugs or food, or may be allergic to the test drug and the related compounds;
* Have a history of severe and uncontrolled diseases, such as cardiovascular, respiratory, gastrointestinal, endocrine, hematologic, mental/nervous systems diseases within one year prior to screening；
* Subjects who have previously undergone surgery that may affect drug absorption, distribution, metabolism, or excretion (e.g., subtotal gastrectomy), or who have a scheduled surgical plan during the study period;
* Use of any DPP-IV enzyme inhibitor within 2 weeks prior to the screening;
* Drug abuse, or positive urine drug screen at screening；
* Smoking more than 5 cigarettes per day within 3 months prior to screening；
* Average alcohol intake is more than 28g alcohol (male) or 14g (female) per week (14g ≈ 497mL beer, or 44mL spirits with low alcohol content, or 145mL wine) within the 3 months prior to screening, or taking any alcohol within 48 hours before dosing, or a positive ethanol breath test at screening；
* Consumption of grapefruit juice, Methylxanthine-rich food or beverage (such as coffee, tea, cola, chocolate, energy drinks) within 48 hours before the administration, or have strenuous exercise, or have other factors affecting drug absorption, distribution, metabolism, excretion, etc.；
* Participation in another clinical trial within 3 months before screening；
* Blood donation (or blood loss) ≥400 mL, or receiving whole blood transfusions or erythrocyte suspension transfusions within 3 months prior to the screening；
* A pregnant/lactating woman, or has a positive pregnancy test at screening or during the trial；
* Estimated glomerular filtration rate (eGFR)<90 mL/min/1.73 m2 calculated by the modification of diet in renal diseases (MDRD) equation at screening；
* Have a positive test result of human immunodeficiency virus (HIV) antibody, or anti-Treponema pallidum specific antibody；
* Currently receiving, or unable to refrain from expected concomitant cytochrome (CYP) 3A inhibitors and inducers;
* Not suitable for this study as judged by the investigator；

Subjects with HI only:

* Drug-induced liver injury；
* Acute liver injury by any cause；
* Subjects with liver failure, or subjects with cirrhosis complicated with hepatocellular carcinoma or symptomatic hepatic encephalopathy, etc., are deemed as unsuitable for this study by the investigator；

Subjects with normal liver function only:

* History of HI, or presence of abnormal results in physical examination and laboratory examination at screening that may indicate any liver illness in the opinion of the Investigator;
* Have a positive test result of hepatitis B surface antigen, or hepatitis C antibody.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2022-05-14 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetic parameters of DBPR108 | Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, and 48 hours after dosing
  Cmax
The pharmacokinetic parameters of DBPR108 | Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, and 48 hours after dosing
  AUC0-t
The pharmacokinetic parameters of DBPR108 | Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, and 48 hours after dosing
  AUC0-inf

SECONDARY OUTCOMES:
The pharmacokinetic parameters of DBPR108 | Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, and 48 hours after dosing
  Tmax
The pharmacokinetic parameters of DBPR108 | Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, and 48 hours after dosing
  t1/2
The pharmacokinetic parameters of DBPR108 | Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, and 48 hours after dosing
  Vz/F
The pharmacokinetic parameters of DBPR108 | Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, and 48 hours after dosing
  CL/F
The number of volunteers with adverse events as a measure of safety and tolerability | Day 1 to Day6
  The number of volunteers with adverse events as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Soochow University, Suzhou, China